CLINICAL TRIAL: NCT03577535
Title: Evaluation of ONCOXIN® in Oral Mucositis, Appetite and Body Mass in Cancer Patients. Real World Setting Study.
Brief Title: Evaluation of ONCOXIN® in Oral Mucositis, Appetite and Body Mass in Cancer Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OOS-CANCER-10
Record Dates: First submitted 2018-06-11; First posted 2018-07-05 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-06

CONDITIONS: Mucositis Oral
Keywords: Oral Mucositis; Nutritional supplement; Chemotherapy; Radiotherapy; Ocoxin / Oncoxin
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oncoxin® (Experimental): Chemo-, radiotherapy or their combination + standard oral mucositis treatment + ONCOXIN
  Interventions: Dietary Supplement: Oncoxin®
- No Oncoxin Treatment® (No Intervention): Chemo-, radiotherapy or their combination + standard oral mucositis treatment.

INTERVENTIONS:
Dietary Supplement: Oncoxin® — Chemo-, radiotherapy or their combination + standard oral mucositis treatment + ONCOXIN 25 ml twice daily for 20 days;
  Arms: Oncoxin®

SUMMARY:
Oral mucositis is one of the most spread side effects of anticancer therapy. It is associated with both chemo- and radiotherapy, decreases QoL, relative dose intensity and leads to nutritive deficiency. Oral mucositis causes secondary infections, increased hospital stay, whereas pain syndrome results in an emotional distress, anorexia and disables natural feeding.

DETAILED DESCRIPTION:
Primary:

To evaluate the efficacy of ONCOXIN on oral mucositis symptoms in patients who receive chemotherapy and/or radiotherapy.

Secondary:

To evaluate the effects of ONCOXIN on nutritional status in patients who receive chemotherapy and/or radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. A signed and dated informed consent form;
2. Patients of both genders, aged 45-75;
3. Malignant neoplasms which have radio-, chemotherapy or their combinations prescribed;
4. ECOG ≤3;
5. WHO oral toxicity scale grade 2 - 3.

Exclusion Criteria:

1. Significant, according to the investigator judgement, concomitant diseases or states which make it complicate or even impossible the patient's participation in the study or make it difficult to interpret the clinical data obtained in any stage of the study always including the following:

   * Mental disorders;
   * Serious/chronic infectious and parasitic diseases;
   * Intolerability to any of ONCOXIN components.
2. Relations with study center personnel (study center staff or family member of the investigator, coordinator or assistant).
3. If the patient fails to assess his/her physical and emotional condition;
4. If the patient fails to comply with the requirements;
5. Patient's refusal to participate in the study;
6. Pregnancy or lactation.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-07-15 (Actual)

PRIMARY OUTCOMES:
Oral mucositis grade in patients during chemotherapy and radiotherapy treatments | 21 days
  Efficacy of OCOXIN on oral mucositis symptoms in patients who receive chemotherapy and/or radiotherapy with WHO oral toxicity scale grades. The WHO scale is dependent on both objective and subjective variables, and measures anatomical, symptomatic as well as functional components of oral mucositis.
  WHO Oral Mucositis Grading Scale:
  * 0 (none): None
  * I (mild): Oral soreness, erythema
  * II (moderate): Oral erythema, ulcers, solid diet tolerated
  * III (severe): Oral ulcers, liquid diet only
  * IV (life-threatening): Oral alimentation impossible

SECONDARY OUTCOMES:
Nutritional status of the patients during Chemotherapy and radiotherapy treatments related with weight gain | 21 days
  Effects of ONCOXIN on nutritional status in patients who receive chemotherapy and/or radiotherapy measured with body mass measures.
Nutritional status of the patients during Chemotherapy and radiotherapy treatments | 21 days
  Effects of ONCOXIN on nutritional status in patients who receive chemotherapy and/or radiotherapy measured with days with the intake of regular food.
Nutritional status of the patients during Chemotherapy and radiotherapy treatments | 21 days
  Effects of ONCOXIN on nutritional status in patients who receive chemotherapy and/or radiotherapy measured with days with no loss of appetite complaints.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Scientific centre of professor Shumsky, Samara, Samara Oblast, Russia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR